CLINICAL TRIAL: NCT02542722
Title: Prevention of Type 2 Diabetes Mellitus (Egabro-Pizarra Study)
Brief Title: Type 2 Diabetes Prevention
Acronym: PIZARRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: Hospital Regional de Malaga (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P09-CTS-5125; PI081592 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2015-05-25; First posted 2015-09-07 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: lifestyle modification; olive oil; Mediterranean diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): General dietary and physical exercise recommendations
  Interventions: Behavioral: Control
- Intervention (Experimental): Intensive intervention on dietary and physical exercise habits.
  Interventions: Behavioral: Intensive Intervention

INTERVENTIONS:
Behavioral: Control — General recommendations about a healthy diet and physical activity and referral to their general physician with a report of the study results in the event of detecting any risk factor or pathological finding
  Arms: Control
Behavioral: Intensive Intervention — Based on office visits each 3 months during the first year, as well as monthly telephone calls during the first year. Each subject will also attend a group educational meeting each 6 months. At each visit they will be given a series of recommendations and their degree of adherence evaluated and the evolution of their weight checked. The recommendations are designed to re-educate the subjects concerning their dietary and physical activity habits
  Arms: Intervention

SUMMARY:
It will be selected 1274 subject older than 40 years of the population of Cabra in order to realize a sociodemographic and habits (toxic, food, of physical activity) survey. It will be realized a physical exploration including anthropometry, blood pressure, oral glucose tolerance test, blood extractions (basal and after 120 ' of the OGTT). Several biochemical determinations will be realized (p.e. marker of fat intake and marker of inflammation) The proposed intervention consists of a series of clinical visits and phone calls programmed with the aim to change the dietetic and physical activity habits of people. The Pizarra study (financed with other grants and realised with the same methodology) will be use as cohort control. Though the basic aim of the project is to achieve a reduction of the of diabetes incidence with a hygienic - sanitary intervention, the ambition of knowing the major number of possible factors that can participate in this process constitutes a complex project capable of analyzing the problem from diverse points of view. Endocrinologists (of two Andalusian hospitals), clinical biochemists, geneticists and dietitians they join in this project to approach an integral way the etiopathogeny of the diabetes type 2.

DETAILED DESCRIPTION:
1. Intervention study population: Egabro Study. This study commenced in 2009 in Cabra, a town of 20,000 inhabitants located in the Subbética region of Cordoba Province (Spain). The study includes persons aged over 40 years.
2. Control population: Pizarra Study. The Pizarra Study is in progress since 1995. The details of this study have been the subject of multiple publications (see CVs). The start of the Egabro Study coincided with the third evaluation of the Pizarra cohort, as well as the extension of the population base, which will now enable the whole population of Pizarra aged over 40 years to be studied.
3. Design: A prospective cohort study with exposure to an intervention on hygiene and health habits:

Cohort A. Egabro Study:

First phase: Cross-sectional prevalence study Second phase: Intensive intervention study in certain risk groups (Cohort study, with a control group)

Cohort B. Pizarra Study:

First phase: Prevalence study (cross-sectional, extension of the initial cohort) Second phase: Follow-up of the cohort, to be used as a control group for the intervention study in the Egabro project 4. Subjects susceptible to the intervention:

1. Persons who, after an oral glucose tolerance test (OGTT), are identified as having the phenotype of Impaired Fasting Glucose (IFG) 2. Persons who, after an OGTT, are identified as having diabetes mellitus. 5. Sampling. Sample size The calculation of the sample size was done according to the recommendations of Carné X et al. (Carné X, et al. Medicina Clín (Barc), 1989; 92:72-73). The sample size was calculated for the main study endpoints based on the Pizarra study data with the aim of decrease the risk of having diabetes about 50% (alpha=0.05, power=90%). The minimum sample size is 479 subject in each cohort. To date, the investigators have enrolled 600 subject each cohort by random sampling.

6. Intervention protocol:

The intervention being undertaken consists of a series of programmed clinical visits and telephone calls in order to change the dietary and lifestyle habits of the participants. Briefly:

Level 1 intervention General recommendations about a healthy diet and physical activity and referral to their general physician with a report of the study results in the event of detecting any risk factor or pathological finding. The procedure is the standard used to date in the Pizarra study and which will continue to be used in this cohort. Subjects with a normal OGTT in the Egabro Study will also be used.

Level 2 intervention

This will consist of an intensive intervention on dietary and physical activity habits as well as Level 1 recommendations. It will be carried out in all those subjects in the Egabro Study who have any alteration after the OGTT: IFG, IGT or previously unknown diabetes. All will be recommended to attend their family physician with a report of the results in order to receive the standard treatment in each case (Level 1 intervention). Additionally, an intervention protocol will be included based on office visits each 4 months during the first year, as well as monthly telephone calls during the first year. Each subject will also attend a group educational meeting each 6 months. At each visit they will be given a series of recommendations and their degree of adherence evaluated and the evolution of their weight checked The recommendations are designed to re-educate the subjects concerning their dietary and physical activity habits:

7.Follow up: two year

SPECIFIC METHODS in basal study and follow up:

Field work (basal and at the end of the first year and second year of the intervention (or observation of the control cohort):

1. An OGTT will be given to all the participants who had an altered OGTT in the baseline study (200 subjects in the Egabro cohort + 200 subjects in the Pizarra cohort).
2. Serum will be obtained fasting and after the OGTT.
3. Records will be made of weight, height, waist and hip circumferences, skinfold thicknesses (suprailiac, subscapular, bicipital and tricipital) and blood pressure.
4. Muscle strength will be estimated as measured by hand grip dynamometry
5. A dietary questionnaire will be given (24 hour recall + frequency survey)
6. An evaluation will be made of physical activity
7. Questions will be asked about any sociodemographic variation and incidence of disease since the previous visit
8. The data will be included in the general database of the project.

Biochemical study (basal and at the end of the first year and second year of the intervention (or observation of the control cohort):

Determination of glucose, insulin, cholesterol, triglycerides, HDL cholesterol, LDL cholesterol, ferritin, C-reactive protein, liver enzymes, urea, uric acid and creatinine in fasting serum and glucose and insulin in post OGTT serum, after one and two year of follow-up.

DATA COLLECTION AND ANALYSIS

1. The first visits have been done by two participating endocrinologists, one registered nurse and one nutritional technician expressly employed for the study (one team in each cohort).
2. Informed consent was requested. Each of the participants completed a questionnaire with closed exhaustive questions. The physical examination was made in accordance with the methods recommended by the WHO (WHO Technical Report Series 854, Geneva 1995). Data were collected on weight, height and waist and hip circumferences of each participant in light clothing and without shoes using a calibrated standardized electronic scale, stadiometer and metric measure. The blood pressure was also taken, with a digital sphygmomanometer (Omron, Hem-703C). The dynamometry was done with the right hand recording three determinations.
3. All the participants, except those who said they were diabetic or who had a capillary blood glucose >180 mg/dL, underwent an OGTT with 75 gr of glucose and venous extraction at baseline and after 2 hours, in accordance with the recommendations of the 1985 WHO technical report. The participants with known or reported diabetes were checked for the diagnosis of diabetes (from the clinical charts) and underwent just fasting blood extraction. Thirty minutes after the extraction the samples are centrifuged "in situ" using a portable centrifuge. The samples are then stored in aliquots and frozen in situ for 15 days before storing them definitively at _80ºC. Determinations are made of blood glucose, cholesterol, HDL cholesterol and triglycerides using routine standardized techniques. The LDL cholesterol is calculated from the Friedewald equation, excluding those participants with triglycerides >400 mg/dL. The blood and serum samples are stored at -80ºC following the protocols of the National DNA Bank for metabolic diseases. The blood is used for genotyping (see below) and the serum for making biochemical and fatty acid measurements (gas chromatography of methyl derivatives) contemplated in the study.
4. The diagnostic criteria for normality, IFG, IGT and type 2 diabetes mellitus used are those established by the 1999 WHO expert committee.
5. The criteria used to define hypertension are those of the US Joint National Committee VI.
6. To typify the weight of the group the body mass index (BMI) is used (BMI = weight in kg/height in m2) and the waist-to-hip ratio. For smoking, participants are considered to be smokers if they smoke or have quit smoking within the previous six months. A family history of type 2 diabetes is considered to be present if the participants report the disease in a first-degree relative (parents, siblings, children).
7. Lipid abnormalities are identified by Brunzell criteria (Brunzell et al. Diabetes Care 2008).
8. Nutritional evaluation: The nutritional questionnaire is designed to collect information about nutritional habits, frequencies and amounts of foods. The following tools are used.

   8.1 Twenty-four hour recall survey: repeated at two different times of the year.

   8.2 Food frequency questionnaire, following the recommendations of Willet (Nutritional Epidemiology. Oxford University Press, Oxford, 1990). The questionnaires are given by experienced dietitians previously trained for this project.

   8.3 The transformation to nutrients of the dietary information is done by computerized conversion according to Moreiras and Martín, modified by one of the researchers of this group using his own sources (Soriguer F. et al. European Journal Epidemiology 13:451-463,1997) as well as other nutrient tables (Mataix J. Universidad de Granada, 2003).

   8.4 Scale of adherence to a Mediterranean diet based on the results of the questionnaires
9. The evaluation of physical activity is done by questionnaires about frequency of activities

ANALYSIS OF THE RESULTS AND STATISTICAL STUDY. All the information derived from the Pizarra and the Egabro studies is collected in specially designed computerized databases. Statistical hypothesis contrast for the variables according to the previsions of the hypothesis elaborated in the design using parametric or non parametric tests according to the adjustment to normality. The strength of the associations in the crosssectional study will be measured by calculating the odds ratio from 2×2 tables or from coefficients of the logistic models when they adjust for possible confounding variables. To compare the incidence / prevention rates of metabolic disorders, the two cohorts will be standardized for age and sex and the relative risks will be calculated with their corresponding CI. The multivariate analysis will be done using Cox regression.

LIMITATIONS: Bias in participation: being a study population, certain groups tend to participate more likely than others. It compensates also working on weekends and holidays to prevent working people participate less. The design is "quasiexperimental". The indication bias of the intervention program carried out will be adjusted using the propensity score method, which enables elimination of the indication bias and making the study closer, using techniques of pairing ("nearest" method) to the most similar situation to that of an experimental study, using probabilities predicted by the logistic models.

Locations:

Local Diabetic Association of Cabra, Córdoba. Local loan from the City Council in Pizarra, Málaga. Research Laboratory Hospital Regional Universitario in Malaga

ELIGIBILITY:
Inclusion Criteria:

* impaired fasting glucose and/or impaired oral glucose tolerance test.

Exclusion Criteria:

* type 2 diabetes mellitus previously diagnosed. In the last 6 months: serious illness or surgery, delivery or breastfeeding.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2009-01; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Incidence of type 2 diabetes in subjects at risk | 12 and 24 months
  Incidence (at 12 and 24 months) of type 2 diabetes diagnosed by oral glucose tolerance test (OGTT) according WHO criteria in subjects with impaired OGTT.

CONTACTS AND LOCATIONS:
Overall Officials: GEMMA ROJO-MARTINEZ, PhD, Study Director — Hospital Regional Universitario de Málaga (Spain)